CLINICAL TRIAL: NCT02575976
Title: Effects of Cardiac Rehabilitation on Functional Capacity and Cardiovascular Risk Factors in Brazilian Patients Assisted by Public Health Care: A Randomized Controlled Trial
Brief Title: Effects of Cardiac Rehabilitation (CR) on Functional Capacity and Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Raquel Rodrigues Britto, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-898235
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Disease; Coronary Disease
Keywords: Rehabilitation; Coronary artery disease; Patient Education; Randomized Controlled Trial; Protocol
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- comprehensive CR (Experimental): education and exercise-based cardiac rehabilitation
  Interventions: Behavioral: comprehensive CR
- exercise-based CR (Active Comparator): Exercise-based cardiac rehabilitation
  Interventions: Other: exercise-based CR
- wait list control (Other): no cardiac rehabilitation
  Interventions: Other: wait list control

INTERVENTIONS:
Behavioral: comprehensive CR — In the comprehensive CR arm, 24 sessions education will be offered, of 30 minutes duration beyond the exercises already performed in the cardiac rehabilitation program (The main program is 6 months in duration, with 36 1-hour exercise sessions)
  Arms: comprehensive CR
Other: exercise-based CR — The main program is 6 months in duration, with 36 1-hour exercise sessions.
  Arms: exercise-based CR
Other: wait list control — No cardiac rehabilitation.
  Arms: wait list control

SUMMARY:
The purpose of this trial are to pragmatically investigate whether participation in a comprehensive CR (i.e., exercise with education) program in a Latin American MIC results in better functional capacity, cardiovascular risk factor control, health behavior, disease-related knowledge, depressive symptoms and lower mortality when compared exercise only CR or wait list control.

DETAILED DESCRIPTION:
The design is a single-blinded, single-site pragmatic superiority RCT with 3 parallel arms: comprehensive CR (education and exercise) versus exercise-based CR (no education, as delivered in Brazil) versus wait list control (i.e., no CR). Patient assessments will be undertaken pre-randomization and again at 6 and 12 months later (in accordance with the end of CR). Mortality will be ascertained at 6 months and 1 year post-recruitment.

The main program is 6 months in duration, with 36 1-hour exercise sessions offered at the following frequencies:

1. participants come to CR for 12 sessions, 3x a week (total of 4 weeks of intervention).
2. participants come to CR for 8 sessions, 2x a week (total of 4 weeks of intervention).
3. participants come to CR for 12 sessions, 1x a week (total of 12 weeks of intervention).

Each participant will receive an individualized exercise prescription based on a grade exercise stress test. Participants will be exercising between 50 and 80% of heart rate reserve. In all stages patients will be requested to exercise in their community other days of the week, to accumulate 30 or more minutes of physical activity at a moderate to vigorous-intensity 5 or more days per week, as recommended in the guidelines.

In the comprehensive CR arm, 24 sessions education will be offered, of 30 minutes duration. More specifically, the education component consists of:

* weekly group education sessions, which are strategically mapped based on patients' information needs and sequenced to support the program learning outcomes. Education sessions are delivered by a health educator team. See table 1 for the CR program schedule, including educational topics (e.g.. diet, medication and exercise).
* A comprehensive education workbook to accompany the sessions, containing 20 chapters. The empirically-validated English version has been translated and culturally-adapted to Brazilian-Portuguese. Clinicians and patients have reviewed the material, and a plain language and clear design review was completed in preparation for this trial.

The standard of care for Brazilian adults with CVD does not include access to CR for all patients, given the gross lack of capacity. All participants will have follow-up appointments with their physician as deemed medically appropriate. Consistent with CONSORT guidelines, usual care will be described in detail for each participant (e.g., number of health visits - both inpatient and outpatient, other treatments).

The number of patients approached and date will be recorded, as well as the reasons for inclusion/exclusion. With informed written consent from the patient and CR clearance from the physician, potentially eligible participants will be scheduled to come on-site to complete pre-test assessments. Participants will be asked to complete a sociodemographic questionnaire, to establish the generalizability of the sample, among other surveys. Clinical information will be extracted from participants' charts.

Eligible participants will be randomized to one of the 3 groups. The randomization sequence was generated using the random.org website in random blocks of 4, with a 1:1:1 allocation ratio. To ensure allocation concealment, the local principal investigator has the allocation sequence in a password-protected file, and will only provide randomization information to the student once it is confirmed the participant is eligible. Due to the nature of the intervention, participants and the doctoral student cannot be blind to treatment allocation.

The primary outcome of functional capacity will be assessed again at 6 months. All other post-test assessments will be undertaken 6 months post-randomization. Mortality will be ascertained from hospital charts and family phone call at 6 months and 1-year. With regard to the baseline and 6 months assessments, participants will be invited to come to the study center to:

1. undertake the shuttle walk test as the indicator of functional capacity,
2. undertake assessments of secondary outcomes including a blood draw for lipids, and
3. complete surveys related to tertiary outcomes.

A master's student blinded to random allocation will undertake post-test assessments, outcome ascertainment and data entry. To minimize loss to follow-up, investigators will send mail and telephone reminders for patients to come on-site for these assessments, based on the Dillman method.

Measures Participants will be asked to complete a sociodemographic questionnaire. Clinical characteristics will be extracted from the medical charts, including sex, age, risk factors, cardiac history, cardiac test results, comorbidities and medications. These are based on the Canadian Cardiovascular Society core element and demographic data definitions. CR session attendance will be extracted from program charts at post-test for participants randomized to the CR arms.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old
* patients living in the Belo Horizonte area

Exclusion Criteria:

* any comorbid physical or serious mental condition which would interfere with the ability to exercise according to CR clinical practice guidelines (i.e., heart failure with ejection fraction less than 45%, complex ventricular dysrhythmia, advanced dementia, leg amputation, advanced cancer, disabling stroke, Parkinson's or substance dependence), and
* any visual or cognitive condition which would preclude the participant from completing the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raquel R Britto, Post doc, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldcroft SA, Taylor NF, Blackstock FC, O'Halloran PD. Psychoeducational rehabilitation for health behavior change in coronary artery disease: a systematic review of controlled trials. J Cardiopulm Rehabil Prev. 2011 Sep-Oct;31(5):273-81. doi: 10.1097/HCR.0b013e318220a7c9. PMID 21734590
- [Background] Dusseldorp E, van Elderen T, Maes S, Meulman J, Kraaij V. A meta-analysis of psychoeduational programs for coronary heart disease patients. Health Psychol. 1999 Sep;18(5):506-19. doi: 10.1037//0278-6133.18.5.506. PMID 10519467
- [Background] Mullen PD, Mains DA, Velez R. A meta-analysis of controlled trials of cardiac patient education. Patient Educ Couns. 1992 Apr;19(2):143-62. doi: 10.1016/0738-3991(92)90194-n. PMID 1299819
- [Background] Schadewaldt V, Schultz T. Nurse-led clinics as an effective service for cardiac patients: results from a systematic review. Int J Evid Based Healthc. 2011 Sep;9(3):199-214. doi: 10.1111/j.1744-1609.2011.00217.x. PMID 21884449
- [Background] Ghisi GL, Abdallah F, Grace SL, Thomas S, Oh P. A systematic review of patient education in cardiac patients: do they increase knowledge and promote health behavior change? Patient Educ Couns. 2014 May;95(2):160-74. doi: 10.1016/j.pec.2014.01.012. Epub 2014 Jan 30. PMID 24529720
- [Background] Chaves GS, Ghisi GL, Grace SL, Oh P, Ribeiro AL, Britto RR. Effects of comprehensive cardiac rehabilitation on functional capacity and cardiovascular risk factors in Brazilians assisted by public health care: protocol for a randomized controlled trial. Braz J Phys Ther. 2016 Nov-Dec;20(6):592-600. doi: 10.1590/bjpt-rbf.2014.0192. Epub 2016 Oct 27. PMID 27849287
- [Background] Herdy AH, Lopez-Jimenez F, Terzic CP, Milani M, Stein R, Carvalho T, Serra S, Araujo CG, Zeballos PC, Anchique CV, Burdiat G, Gonzalez K, Gonzalez G, Fernandez R, Santibanez C, Rodriguez-Escudero JP, Ilarraza-Lomeli H. South American guidelines for cardiovascular disease prevention and rehabilitation. Arq Bras Cardiol. 2014 Aug;103(2 Suppl 1):1-31. doi: 10.5935/abc.2014s003. No abstract available. English, Portuguese. PMID 25387466
- [Background] Grace SL, Turk-Adawi KI, Contractor A, Atrey A, Campbell NR, Derman W, Ghisi GL, Sarkar BK, Yeo TJ, Lopez-Jimenez F, Buckley J, Hu D, Sarrafzadegan N. Cardiac Rehabilitation Delivery Model for Low-Resource Settings: An International Council of Cardiovascular Prevention and Rehabilitation Consensus Statement. Prog Cardiovasc Dis. 2016 Nov-Dec;59(3):303-322. doi: 10.1016/j.pcad.2016.08.004. Epub 2016 Aug 17. PMID 27542575
- [Result] Chaves GSDS, Ghisi GLM, Grace SL, Oh P, Ribeiro AL, Britto RR. Effects of comprehensive cardiac rehabilitation on functional capacity in a middle-income country: a randomised controlled trial. Heart. 2019 Mar;105(5):406-413. doi: 10.1136/heartjnl-2018-313632. Epub 2018 Oct 3. PMID 30282639
- [Result] Chaves GSS, Lima de Melo Ghisi G, Britto RR, Grace SL. Maintenance of Gains, Morbidity, and Mortality at 1 Year Following Cardiac Rehabilitation in a Middle-Income Country: A Wait-List Control Crossover Trial. J Am Heart Assoc. 2019 Feb 19;8(4):e011228. doi: 10.1161/JAHA.118.011228. PMID 30764702
- [Derived] Ghisi GLM, Chaves GSS, Ribeiro AL, Oh P, Britto RR, Grace SL. Comprehensive Cardiac Rehabilitation Effectiveness in a Middle-Income Setting: A RANDOMIZED CONTROLLED TRIAL. J Cardiopulm Rehabil Prev. 2020 Nov;40(6):399-406. doi: 10.1097/HCR.0000000000000512. PMID 32694454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
Started | 37 | 39 | 39
Completed | 32 | 31 | 30
Not Completed | 5 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control | Total
Number analyzed (Participants) | 37 | 39 | 39 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.8) | 59.0 (9.9) | 58.7 (9.6) | 59.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 33
  Male | 27 | 28 | 27 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Low Education [Count of Participants; unit: Participants] — It was considered low education those participants who did not complete high school.
  Participants | 21 | 33 | 28 | 82
Marital status - Married [Count of Participants; unit: Participants] | 20 | 27 | 27 | 74
Work status - employed [Count of Participants; unit: Participants] | 15 | 14 | 17 | 46
Low Monthly income [Count of Participants; unit: Participants] — It was considered low monthly income those participants who receive less than four minimum wages per month.
  Participants | 31 | 34 | 35 | 100

OUTCOME MEASURES:

1. Primary Outcome: Functional Capacity Assessed by Changes in Total Distance Walked in the Incremental Shuttle Walk Test
Description: The Incremental Shuttle Walk Test (ISWT). The ISWT consists of an incremental, walking test where participants are required to walk up and down a 10-meter course. The speed of walking, which is increased by a small increment every minute (0.17 ms-l), is externally paced and controlled by audio signals played from a tape recorder19. There are 12 levels in total, beginning with 0.5 ms-1, and each level lasts for one minute. At the end of each minute, exercise heart rate (HR) and rating of perceived exertion (RPE) scores will be recorded. For this test, the higher the number of meters, the higher the functional capacity.
Time Frame: Functional capacity measured by walked distance in the ISWT at 6 months
Population: The analyzed population was based on the threshold sessions: a minimum of 24 exercise sessions and 16 education classes. The presented results considered the Per Protocol analysis, explaining the different numbers in the flow diagram and the analyzed numbers.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
Number analyzed (Participants) | 26 | 25 | 30
meters | 488.1 (106.3) | 464.8 (121.6) | 394.0 (171.9)

2. Secondary Outcome: Risk Factors Measurement of Systolic Blood Pressure
Description: Blood pressure was assessed using the validated 7670-06 mobile stand (Welch Allyn Inc., Skaneateles Falls, NY, USA). Mean systolic blood pressure value was recorded, and hypertension was considered where values exceed 140/90 mmHg and/or participant was taking a blood pressure-lowering medication
Time Frame: Systolic blood pressure measured at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
Number analyzed (Participants) | 26 | 25 | 30
mmHg | 114.6 (19.2) | 114.4 (16.3) | 120.0 (18.4)

3. Secondary Outcome: Risk Factors Measurement of Waist Circumference.
Description: Waist circumference was assessed at the superior border of the iliac crest. Values greater than 102 cm in men and 88 cm in women were considered indicative of central obesity.
Time Frame: Waist circumference measured at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
Number analyzed (Participants) | 25 | 24 | 28
centimeters | 95.5 (13.4) | 93.0 (10.0) | 94.9 (9.4)

4. Secondary Outcome: Risk Factors Measurement of Fasting Blood Glucose Values
Description: Fasting blood glucose values were extracted from center charts. Dysglycemia was considered present where fasting blood glucose exceeded 126 mg/dl and/or participant was taking a glucose-lowering medication
Time Frame: Glycaemia measured at 6 months
Population: The analyzed population was based on the threshold sessions: a minimum of 24 exercise sessions and 16 education classes. The presented results considered the Per Protocol analysis, explaining the different numbers in the flow diagram and the analyzed numbers. Sample size reduced because difficult to obtain the results in a reasonable time frame.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
Number analyzed (Participants) | 6 | 5 | 6
mg/dl | 99.8 (20.9) | 98.8 (27.3) | 94.2 (10.4)

5. Secondary Outcome: Risk Factors Measurement of Total Cholesterol Values.
Description: Total cholesterol values were extracted from center charts and dyslipidemia was considered present where total cholesterol values exceeded 240 mg/dl and/or participant was on a lipid-lowering agent.
Time Frame: Cholesterol measured at 6 months.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
Number analyzed (Participants) | 7 | 7 | 7
mg/dl | 150.6 (25.4) | 169.3 (51.0) | 153.1 (29.8)

6. Other Pre Specified Outcome: Heart-health Behaviors
Description: Assessed by questionnaires.
Time Frame: Measured at 6 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Comprehensive CR | Exercise-based CR | Wait List Control
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/39 | 1/39
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02575976/Prot_SAP_000.pdf